CLINICAL TRIAL: NCT06946459
Title: Effects of Hip Strength Exercise Training on Jump Distance, Hip Muscle Strength and Throwing Performance in 15-19-Year-Old Female Handball Players
Brief Title: Impact of Hip Strength Training on Jump and Throw Performance in Young Female Handball Players
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Zümre Hediye TAŞÇI, MSc Student, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IstanbulU-SportsMed-ZHT-01
Record Dates: First submitted 2025-04-19; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Strength Training Effects
Keywords: Handball players; Strength training effects; Throwing performance; Jumping performance
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: In our study, the athletes were randomly assigned to two groups: the Hip Strength Exercise Training Group and the Control Group. The Hip Strength Exercise Training Group consists of handball players who were planned to receive hip strength exercise training three times a week for 8 weeks following the initial assessments. The Control Group, on the other hand, represents handball players who were instructed to continue with their regular handball training for 8 weeks after the initial assessments.
Who Masked: Outcomes Assessor
Masking Description: In this study, the participants were not blinded to their group assignment, as it was evident which group they belonged to (Hip Strength Exercise Training Group or Control Group) based on the intervention. However, the outcomes assessors were blinded to group allocation to reduce potential bias in the measurement of the outcomes. This masking ensured that the evaluation of the effects of the intervention remained unbiased.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hip Strength Exercise Training Group (Experimental): This group received a hip strength exercise training program in addition to their regular handball training for 8 weeks, three sessions per week. The intervention aimed to improve hip muscle strength, jump distance, and throwing performance.
  Interventions: Other: Exercise
- Control Group (No Intervention): This group continued their regular handball training without any additional intervention during the 8-week study period. They served as the control group to compare the effects of the hip strength exercise training.

INTERVENTIONS:
Other: Exercise — Participants in the Hip Strength Exercise Training group performed structured hip strengthening exercises using resistance bands in addition to their regular handball and strength training programs. The training was implemented three times per week for 8 weeks, with one rest day between sessions, and was conducted before regular handball practices. The exercises focused on activating and strengthening the hip muscles through simple, well-structured movements. Resistance bands were chosen due to their portability, cost-effectiveness, and suitability for adolescent athletes. This method ensured a safe training environment, reduced the risk of overload, and allowed for proper execution and control of the exercises.
  Arms: Hip Strength Exercise Training Group

SUMMARY:
This study aims to investigate the effects of an 8-week Hip Strength Exercise Training program, implemented in addition to the athletes' regular training routines, on hip muscle strength, jump distance, and three-step jump shot performance in female handball players aged 15 to 19. Furthermore, the study seeks to explore the potential relationships between throwing performance and various physical parameters, including anthropometric measurements, handgrip strength, and body fat percentage.

DETAILED DESCRIPTION:
Handball is a complex and multifactorial team sport determined not only by each player's individual performance but also by the tactical components and interactions within the team. Therefore, defining the game and identifying the key factors influencing performance remain challenging. Handball players must effectively coordinate basic motor skills such as running, jumping, pushing, and changing direction, along with handball-specific skills like passing, catching, controlling, and blocking, to execute shots or create optimal scoring opportunities for teammates.

Since the winning team in handball is the one that scores the most goals, goal shooting is one of the most critical aspects of the game. A successful goal shot requires the ball to reach maximum velocity and be accurate enough to deceive the goalkeeper. The faster and more accurately the ball is thrown, the less time defenders and the goalkeeper have to react and intervene.

In addition to throwing speed and accuracy, jump distance is also a significant factor influencing performance in handball matches. The most frequently used shot type in handball competitions is the jump shot. The energy produced during a jump shot originates from the force exerted against the ground. The higher the player jumps, the longer the flight time, increasing the likelihood of avoiding defensive blocks.

Handball demands high levels of explosive strength, maximal strength, and muscular power in both the upper and lower extremities. While training programs are generally multidimensional, it is important to identify which muscle groups contribute most significantly to performance in order to optimize training approaches. This is because many handball-specific skills such as throwing, blocking, pushing, and holding require considerable strength and power output.

The hip plays a critical role in handball shooting by initiating upper body movement and transferring momentum from the lower to the upper extremities. It provides a stable base for the upper body during the shot, thereby playing a significant role in shot performance. Well-designed hip strengthening programs have been shown to yield not only improvements in strength but also positive effects on secondary outcomes such as linear sprinting, agility, change of direction, and sport-specific performance metrics.

The existing literature highlights a lack of sufficient research examining the relationship between physical capacity and throwing performance. There is a particular need for studies investigating the effects of muscle strength, jump distance, and overall physical fitness on throwing performance. Moreover, it has been noted that studies focusing on female handball players are relatively limited compared to those involving males, underscoring the need for further research in this area.

In this thesis study, we aim to investigate the effects of an 8-week Hip Strength Exercise Training program, implemented in addition to routine training, on hip muscle strength, jump distance, and three-step jump shot performance in female handball players aged 15 to 19. Additionally, we aim to examine the relationships between throwing performance and anthropometric measurements, handgrip strength, and body fat percentage.

We hypothesize that the Hip Strength Exercise Training program will positively contribute to throwing performance by improving hip muscle strength, throwing speed, throwing accuracy, and jump distance. Accordingly, we suggest that low-cost, easily applicable hip strengthening exercises utilizing resistance bands can be integrated into training routines and contribute to the development of injury prevention strategies.

Based on the above, our hypotheses are as follows:

Hypothesis 1: Hip Strength Exercise Training in handball players has a positive effect on hip muscle strength.

Hypothesis 2: Hip Strength Exercise Training in handball players has a positive effect on throwing accuracy.

Hypothesis 3: Hip Strength Exercise Training in handball players has a positive effect on throwing speed.

Hypothesis 4: Hip Strength Exercise Training in handball players has a positive effect on jump distance.

ELIGIBILITY:
Inclusion Criteria:

* Signing the Informed Voluntary Consent Form by agreeing to voluntarily participate in the study
* Being a handball player aged between 15-19 years
* Being female
* Having reached menarche
* Having the ability to understand and speak

Exclusion Criteria:

* Having sustained an extremity injury in the last 6 months
* Having a body mass index (BMI) greater than 25 kg/m² (obesity)
* Having a cardiovascular, neurological, or pulmonary disease
* Experiencing hip pain related to loading and fatigue, or hip pain due to muscle and spasms
* Presence of bursitis, synovitis, arthritis, or osteomyelitis in the hip

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — The study includes female handball players .
Enrollment: 34 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-02-23 (Actual); Study Completion 2025-04-27 (Estimated)

PRIMARY OUTCOMES:
Throwing Velocity | two weeks, baseline and after 8-week intervention period
  Throwing velocity was measured using the Doppler radar gun (Bushnell Speedster III). Participants performed jump shots from behind the 9-meter line using the three-step technique. The average ball speed (km/h) from five valid throws to each corner of the goal was recorded. The radar gun was placed 4 meters behind the free throw line and aligned with the release height and target corner to ensure measurement accuracy.
Throwing Accuracy | two weeks, baseline and after 8-week intervention period
  Throwing accuracy was evaluated by targeting 50 cm circular zones placed in the upper right, upper left, and lower corners of a standard handball goal. Five throws per corner were completed, and the number of successful throws passing through the designated target area was recorded.

SECONDARY OUTCOMES:
Anthropometric Measurements | one weeks, baseline
  Circumference and length measurements (shoulder, upper arm, forearm, wrist, arm span, etc.) will be performed according to International Society for the Advancement of Kinanthropometry protocols using flexible fabric measuring tapes.
Body Fat Percentage | one weeks, baseline
  Body fat percentage will be assessed using the bioelectrical impedance analysis device (Tanita TBF-300 M).
Hand Grip Strength | one weeks, baseline
  Hand grip strength will be measured using the hydraulic hand dynamometer (Jamar), assessing the overall strength of the participant's hand muscles.
Countermovement Jump Distance | two weeks, baseline and after 8-week intervention period
  Vertical jump performance will be evaluated through the modified counter movement jump test, measured using a digital jump meter (Takei), to assess explosive lower-body power.
Single Leg Vertical Jump (SLVJ) Distance | two weeks, baseline and after 8-week intervention period
  Vertical jump distance on the dominant leg will be measured using a digital jump meter (Takei) to assess unilateral leg power.
Single Leg Horizontal Jump (SLHJ) Distance | two weeks, baseline and after 8-week intervention period
  Horizontal jump distance on the dominant leg will be evaluated using a flat measurement tape fixed to the ground to assess functional leg strength and coordination.
Hip Muscle Strength | two weeks, baseline and after 8-week intervention period
  Hip concentric extension and flexion strength and endurance will be measured using the isokinetic device (Cybex Humac Norm). The tests will involve 4 maximum concentric contractions for strength and 15 for endurance at 180°/s speed, following 5 practice trials.

CONTACTS AND LOCATIONS:
Overall Officials: Zümre H Taşçı, MSc student, Principal Investigator — Istanbul University; Sertaç Yakal, Dr., Principal Investigator — Istanbul University
Locations (1):
- Department of Sports Medicine Istanbul Unıversıty, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No